CLINICAL TRIAL: NCT03294395
Title: New Antibiotic Treatment Options for Uncomplicated Anogenital Gonorrhoea Infections - a Double-blind Randomized Controlled Non-inferiority Trial
Brief Title: New AntiBiotic Treatment Options for Uncomplicated Anogenital GOnorrhoea
Acronym: NABOGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Public Health Service of Amsterdam (Other Government)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Henry J.C. de Vries, Professor MD, PhD, Public Health Service of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NABOGO
Record Dates: First submitted 2017-09-18; First posted 2017-09-27 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Gonorrhea
Keywords: Antimicrobial resistance; Antibiotics; Fosfomycin; Ertapenem; Gentamicin; Neisseria Gonorrhoeae
MeSH Terms: conditions — Gonorrhea | interventions — Ertapenem; Fosfomycin; Gentamicins; Injections; Ceftriaxone

STUDY DESIGN:
Intervention Model Description: A double-blind randomized clinical trial with non-inferiority design
  *since October 2018 one study arm (fosfomycin) has been dropped. In a subset of these participants the plasma concentration of ceftriaxone, ertapenem and gentamicin is measured.
  An open-label randomized substudy evaluating the pharmacokinetics of ceftriaxone ertapenem and fosfomycin in 60 healthy volunteers (this number is in addition to the 346 NABOGO participants with gonorrhea)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants receive either intramuscular treatment and if applicable intramuscular placebo. Both particpant and care provider are blind to the regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ceftriaxone im (Active Comparator): Current standard treatment. Ceftriaxone 500mg (single intramuscular dose) + placebo (single oral dose)
  Interventions: Drug: Ceftriaxone
- Ertapenem im (Experimental): Ertapenem 1000mg (single intramuscular dose) + placebo (single oral dose)
  Interventions: Drug: Ertapenem 1000 MG
- Fosfomycin po (Experimental): Fosfomycin oral suspension 6g (single oral dose) + placebo (single intramuscular dose)
  Interventions: Drug: Fosfomycin Oral Suspension
- Gentamicin im (Experimental): Gentamicin sulfate, injectable 5mg/kg (single intramuscular dose) + placebo (single oral dose)
  Interventions: Drug: Gentamicin Sulfate, Injectable

INTERVENTIONS:
Drug: Ertapenem 1000 MG — single dose 1000mg intramuscular injection
  Other Names: Invanz
  Arms: Ertapenem im
Drug: Fosfomycin Oral Suspension — single dose 6g oral suspension
  Other Names: Monuril
  Arms: Fosfomycin po
Drug: Gentamicin Sulfate, Injectable — single dose 5mg/kg (maximum 400mg) intramuscular injection
  Other Names: no other names
  Arms: Gentamicin im
Drug: Ceftriaxone — single dose 500mg intramuscular injection
  Other Names: no other names
  Arms: Ceftriaxone im

SUMMARY:
This study evaluates the efficacy of three experimental antibiotics in the treatment of uncomplicated anogenital gonorrhoea. Participants will be randomized to one of four study arms and will receive either one of the three experimental antibiotics (ertapenem, fosfomycin and gentamicin) or the current standard antibiotic (ceftriaxone). Both the study team and the participant are blinded to the administered treatment. This enables the investigators to compare the eradication capacity and safety of the experimental antibiotics with the standard treatment.

*Following the advise of the DSMB based on a planned interim analysis, in October 2018 one study arm (fosfomycin 6g PO) was dropped and the randomized clinical trial was continued with three treatment arms (ceftriaxone 500mg IM, ertapenem 1000mg IM and gentamicin 5mg/kg IM) and without the oral placebo.

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) to extended spectrum cephalosporins (ESC) among Neisseria gonorrhoeae (Ng) is a major public health concern. With no alternative antimicrobial treatment options for gonorrhoea and only a few new drugs in the development pipeline, it is important to test existing antibiotics for their efficacy in gonorrhoea treatment. This project aims to identify new treatment modalities for uncomplicated gonorrhoea using the registered drugs ertapenem, fosfomycin and gentamicin. This trial is a double blind randomized clinical non-inferiority trial with four treatment arms. 108 participants are randomly assigned to each study arm . Participants will receive either ceftriaxone 500mg intramuscularly (IM) or ertapenem 1000mg IM or gentamicin 5mg/kg IM with a maximum of 400mg (in two doses) supplemented with an oral placebo, or receive fosfomycin 6g oral suspension supplemented with an intramuscular placebo. The bacterial eradication capacity of the study antimicrobials at the included infection site is measured 7-14 days after treatment, using an RNA-based Nucleic Acid Amplification Test (NAAT).

*Following the advise of the DSMB based on a planned interim analysis, in October 2018 one study arm (fosfomycin 6g PO) was dropped and the randomized clinical trial was continued with three treatment arms (ceftriaxone 500mg IM, ertapenem 1000mg IM and gentamicin 5mg/kg IM) and without the oral placebo.

ELIGIBILITY:
Inclusion criteria main study

* 18 years or older
* Anorectal, cervical/vaginal or urethral Ng infection, diagnosed by the following:

  * Ng-positive Gram-stained smear (intracellular Gram-negative diplococci and leukocytes) and/or
  * Positive for Ng by nucleic acid amplification test (NAAT) (Aptima Combo 2) and/or
  * Positive for Ng by culture
* Provide samples from the included infection site for NAAT and direct culture immediately before treatment
* Willing to abstain from anal, vaginal and oral sex until the test of cure (TOC)-visit, or use condoms during sex
* Willing and able to return for a TOC-visit 7-14 days after treatment
* Provide informed consent
* Accept intramuscular injections

Exclusion criteria main study

Pre-randomisation:

* Suspicion of a complicated Ng infection based on signs and/or symptoms indicating pelvic inflammatory disease (PID), epididymitis, prostatitis or gonococcal arthritis*
* Another (sexually transmitted) infection or a suspicion of another infection for which systemic antimicrobial therapy is indicated
* Pregnancy, having a wish to become pregnant or breastfeeding (tested at inclusion visit)
* Not able to read/understand Dutch or English
* HIV infection if:

  * Newly diagnosed HIV infection (upon the inclusion visit) and/or
  * CD4+ cell-count <200 cells/μL (as reported by the patient)
* Known allergy or adverse reactions to ceftriaxone, ertapenemor gentamicin
* Known renal impairment (based on estimated GFR using Cockroft and Gault formula using serum creatinin measured with a point-of-care (POC) test; cut off value renal impairment eGFR ≤ 50 ml/min)
* Known liver cirrhosis (based on history)
* Known congestive heart failure (based on history)
* Known myasthenia gravis
* Known hearing loss or balance disorder, confirmed by an ear-nose-throat (ENT)-doctor or for which an ENT doctor has been consulted and a diagnostic process is still in progress (based on history)
* Concurrent use of any of the following medication:

  * systemic antibacterial antimicrobials other than nitrofurantoin or metronidazole
  * systemic immunosuppressive drugs
  * systemic valproic acid
* Use of any antimicrobial therapy other than nitrofurantoin or metronidazole in the two weeks prior to study enrollment (based on history)
* Previous enrollment in the study
* Concurrent participation in other non-observational medical research*
* Unlikely to adhere to the study protocol

Post-randomisation:

Exclusion of participants from the modified intention to treat analysis (mITT):

* Negative result of Ng NAAT of sample collected on T0 (the day of treatment). This could be the case in the following situations:

  1. Negative NAAT in spite of positive gram stain.
  2. Positive NAAT on pre-study visit but spontaneous clearance of the infection in the time period between first test and return visit for treatment (=study inclusion visit). A novel sample for NAAT will be collected on the study inclusion visit just before administration of treatment; if these results are Ng-negative a participant will be excluded of mITT.
* Loss to follow-up, i.e. no study visit TOC 7-14 days after treatment administration.

Exclusion from per protocol analysis (PP):

* Exclusion of mITT
* Use of non-study related antibiotics after inclusion and prior to TOC visit
* Condomless sexual contact with the primary anatomical gonorrhea site involved after inclusion and prior to TOC visit
* Other protocol violations

Inclusion criteria PK substudy (healthy volunteers):

* 18 years or older
* Provide informed consent

Exclusion criteria PK substudy (healthy volunteers)

Pre-randomisation:

* Pregnancy, having a wish to become pregnant or breastfeeding (tested at inclusion visit)
* Not able to read/understand Dutch or English
* Known allergy or adverse reactions to ceftriaxone, ertapenem, or fosfomycin.
* Known renal impairment (based on estimated GFR using Cockroft and Gault formula using serum creatinin measured with a point-of-care (POC) test; cut off value renal impairment eGFR ≤ 50 ml/min)
* Known liver cirrhosis (based on history)
* Concurrent use of any of the following medication:

  * systemic valproic acid
  * systemic metoclopramide
* Use of any systemic antimicrobial therapy other than nitrofurantoin or metronidazole in the two weeks prior to study enrollment (based on history)
* Concurrent participation in other non-observational medical research (apart from NABOGO RCT)
* Unlikely to adhere to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with treatment success in each study arm for the included anatomic infection | 7-14 days after treatment
  Proportion of participants with treatment success in each study arm using a molecular test (Nucleic acid amplification test, NAAT). Treatment succes is defined as a negative test of cure (NAAT) 7-14 days after treatment.

SECONDARY OUTCOMES:
Proportion of participants with treatment success in each study arm at all anatomical infection sites | 7-28 days after treatment
  Proportion of participants with treatment success in each study arm using a molecular test (Nucleic acid amplification test, NAAT). Treatment succes is defined as a negative test of cure (NAAT) 7-28 days after treatment.
Incidence of treatment-emergent adverse events | until 30 days after treatment
  The incidence, type and severity of treatment-related adverse events as assessed by CTCAE v4.0 will be measured.
Antimicrobial susceptibility of Ng-strains to study antibiotics | Day 0 (before treatment) - 28 (after treatment)
  The in vitro antimicrobial susceptibility (in MIC) of the experimental and reference treatment will be measured in all Ng strains collected at all infected anatomical sites of each participant at inclusion and in case of a positive test of cure.
Blood plasma concentration of ceftriaxone, ertapenem and gentamicin in a subset of 60 NABOGO participants | within 24 hours after treatment administration
  The blood plasma concentration will be measured 1 times within the first 24 hours after treatment administration. With these measurements the investigators will estimate the population pharmacokinetics of ceftriaxone, ertapenem and gentamicin.
Duration of symptoms after treatment | 1-30 days after treatment
  All participants are asked to report their symptoms daily in a diary, this will be evaluated at the follow-up visit (7-14 days after treatment) and at the online evaluation questionnaire (30 days after treatment). The mean duration of all symptoms after treatment will be measured for all study antibiotics.
Clinical and demographic predictors for treatment failure | until 7-14 days after treatment
  The investigators will measure if demographic (e.g. gender, HIV status) and clinical factors (e.g. anatomical location, duration of symptoms before treatment) are associated with treatment failure (treatment failure is defined as any case in which the participant received escape medication).
Blood plasma concentration of ceftriaxone, ertapenem and fosfomycin in 60 healthy volunteers | 24 hours
  Healthy volunteers will be randomly assigned to one of the three antibiotics. After administration of the antibiotic, the blood plasma concentration will be measured 4 times within the first 24 hours. With these measurements the investigators will estimate the population pharmacokinetics of ceftriaxone, ertapenem and fosfomycin.

CONTACTS AND LOCATIONS:
Overall Officials: Henry JC de Vries, PhD, MD, Principal Investigator — Public Health Service of Amsterdam
Locations (1):
- Public Health Service, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Teker B, Schim van der Loeff M, Boyd A, Mathot R, van Dam A, de Vries H, Jongen VW. Diarrhoea as a frequent adverse event after intramuscular ertapenem treatment for uncomplicated Neisseria gonorrhoeae: a secondary analysis from the NABOGO trial. Sex Transm Infect. 2026 Jan 16:sextrans-2025-056735. doi: 10.1136/sextrans-2025-056735. Online ahead of print. PMID 41545057
- [Derived] Teker B, de Vries H, Heijman T, van Dam A, Schim van der Loeff M, Jongen VW. Spontaneous clearance of asymptomatic anogenital and pharyngeal Neisseria gonorrhoeae: a secondary analysis from the NABOGO trial. Sex Transm Infect. 2023 Jun;99(4):219-225. doi: 10.1136/sextrans-2022-055488. Epub 2022 Jul 12. PMID 35820778
- [Derived] de Vries HJC, de Laat M, Jongen VW, Heijman T, Wind CM, Boyd A, de Korne-Elenbaas J, van Dam AP, Schim van der Loeff MF; NABOGO steering group. Efficacy of ertapenem, gentamicin, fosfomycin, and ceftriaxone for the treatment of anogenital gonorrhoea (NABOGO): a randomised, non-inferiority trial. Lancet Infect Dis. 2022 May;22(5):706-717. doi: 10.1016/S1473-3099(21)00625-3. Epub 2022 Jan 19. PMID 35065063

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Initial version (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT03294395/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Last Amended version (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03294395/Prot_SAP_001.pdf